CLINICAL TRIAL: NCT03397940
Title: Investigating the Role of Structured Days on Accelerated Weight Gain During Summer: A Natural Experiment
Brief Title: Role of Structured Days on Weight Gain
Status: Completed | Type: Observational
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, R. Glenn Weaver, Assistant Professor, University of South Carolina
Other Study IDs: Pro00065211
Record Dates: First submitted 2017-11-10; First posted 2018-01-12 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Body Weight; Cardio-respiratory Fitness; Sleep; Nutrition Poor; Physical Activity; Screen Time
MeSH Terms: conditions — Body Weight; Malnutrition; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Year Round School: Children attending year round school
- Traditional School: Children attending a traditional school with a traditional calendar school year

SUMMARY:
Summer vacation is a 3-month window of vulnerability for children from low-income households when health behaviors and academic learning decay. The goal of this project is to collect information on where low-income children go during summer, what they do when they get there, and how their behaviors (physical activity, sedentary, sleep, and diet) differ between the summer (unstructured days) and school year (structured days). This study is 1) significant because it will provide evidence on potential points of intervention that can reduce or reverse the excessive unhealthy weight gains that occur during summer and 2) innovative because it will be the first to identify changes in activity, sedentary, sleep, and dietary behaviors during prolonged and shorter periodic breaks from school and link these behaviors to changes in zBMI over time.

DETAILED DESCRIPTION:
For children (5-12yrs) from low-income households, summer vacation is a "window of vulnerability" and represents an extended period of time (typically 9-10 weeks) in which declines in academic performance occur. For 30 years, empirical evidence has indicated that children from low-income households experience greater declines in reading and math skills during the summer vacation than their middle-to-upper income peers. Additionally, a growing body of evidence demonstrates that the amount of weight gained during summer vacation is 3-5 times greater than the amount of weight gained during the school year. Moreover, this excessive weight gain during summer is more pronounced for low-income, minority children, the same children experiencing the greatest summer learning loss. What children eat and drink, the types of physical activity opportunities, and the amount of screen-time and sleep (two important correlates of weight gain) they engage in during summer vacation is unknown. However, a substantial body of literature indicates that children engage in a greater number of obesogenic behaviors during less-structured times (e.g., weekend days) compared to more-structured times (e.g., week/school days). This phenomenon is refered to as the Structured Days Hypothesis. These behaviors include 1) increased time spent sedentary, 2) reduced engagement in physical activity, 3) displaced sleep patterns, and 4) unhealthy dietary patterns. This study hypothesizes that summer vacation is simply one long weekend where the effect of children's obesogenic behaviors on weight are compounded over a three month time period. However, should children be involved in a structured program over the summer they would not engage in obesogenic behaviors and they would not experience unhealthy weight gains and fitness loss. Recently, one school district in the Columbia, SC area adopted a year-round calendar for an elementary school. This provides a unique opportunity to conduct a natural experiment examining the effects of shorter periodic breaks vs. one prolonged break from structured days (i.e., school days) on the obesogenic behaviors, weight gain, and fitness. This study will use a two arm accelerated longitudinal cohort design to complete the following specific aims: Aim 1: Compare changes in BMI z-scores and fitness during the traditional 3-month summer and 9-month school year between children attending a school that follows a year-round school calendar to children attending match-paired schools that follow a traditional school calendar. Aim 2: Compare changes in sleep, physical activity, sedentary behaviors, and diet during the traditional 3-month summer and 9-month school year between children attending a school that follows a year-round school calendar to children attending match-paired schools that follow a traditional school calendar. This study is significant because the reason for children's weight gain and fitness loss during the summer is unknown. This study is innovative because no studies have examined the effects of prolonged (9 weeks all at once) vs. periodic breaks (3 week breaks distributed throughout the year) from a structured environment on children's weight and fitness.

ELIGIBILITY:
Inclusion Criteria:

K, 1st, 2nd, and 3rd grade students without any physical and/or medical conditions that would limit their ability to take part in measurements.

Exclusion Criteria:

Children in the 4th and 5th grade will be excluded from participation in the obesogenic behavior assessments because they will move out of elementary school over the two-year study.

Ages: 5 Years to 9 Years | Sex: All
Age Groups: Child
Study Population: Three schools (2 traditional and 1 year-round) enrolling 1,279 students have agreed to participate. 85.0% of children in these schools qualify for free and/or reduced price lunch, and 67.5% of children attending these schools are black, 28.5% are white, and 3.6% are Hispanic. The first school was selected to participate because it operates on a year-round calendar. The second and third schools were selected because their enrollment size and student demographics closely match the enrollment and student demographics of the first school. All children in the participating schools will have their height/weight and cardiovascular fitness measured.
Sampling Method: Probability Sample
Enrollment: 2279 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | Baseline and will follow up at 4 months, 12 months, 16 months, and 24 months
  All students enrolled in the partnering schools will have their height and weight measured using standard procedures, as part of their routine PE class. Height and weight will be collected prior to and following every break lasting 3 weeks or longer. These measures will be collected with the help of trained research staff during regularly scheduled PE classes to ensure data quality. This information will be used to compare the BMI (translated into age/sex z-scores [zBMI] for analytical modeling) over time and between students attending a year-round school and traditional schools. These tests are valid and reliable for this age group.
Change in Cardiorespiratory Fitness: | Baseline and will follow up at 4 months, 12 months, 16 months, and 24 months
  All students enrolled in the partnering schools will take part in the cardiovascular fitness (CVF) test (i.e., PACER) as part of their routine PE class. These tests are administered to this age group and occur as part of regular PE class as part of a South Carolina statewide assessment system.This information will be used to compare the CVF over time and between students attending a year-round school and traditional schools. These tests are valid and reliable for this age group.

SECONDARY OUTCOMES:
Change in Sleep | Baseline and follow up at 3 months, 12 months, and 15 months
  Children's sleep will be assessed via wrist-placed Actigraph Links.
Change in Dietary Behavior | Baseline and follow up at 3 months, 12 months, and 15 months
  Dietary patterns rather than individual foods will be assessed. For the current study, the intent is to estimate less healthful/more healthful foods and beverages consumed and compare these between summer and school. The study will assess child dietary patterns using two approaches. First, a modified dietary screener questionnaire will be completed by a parent/guardian at each measurement (traditional school and summer vacation) each year. Screener items were selected from multiple screeners developed for use in this age group and have been widely used in research. The screeners are the 26-item Dietary Screener Questionnaire,16 items from the National Youth Physical Activity and Nutrition Study, and items from several additional food/beverage validated screeners. These dietary screeners provide accurate estimates of food groups and dietary patterns, to allow for examination of relationships between diet and other variables in this study. These screeners have been tested for validity
Change in Physical Activity | Baseline and follow up at 3 months, 12 months, and 15 months
  Time (minutes per day) spent sedentary, and in light, moderate, and vigorous physical activity will be collected using a non-dominant wrist-placed ActiGraph Link for 9-days (common timeframe to collect physical activity data). Non-dominant wrist-placement provides an advantage over waist placement by improving compliance and the ability to collect information regarding sleep. The device is water-proof, allowing us to capture water activities during summer. A calibration/validation study was recently published to establish methodology to distill activity-intensities from wrist-placed ActiGraph in children. The widely accepted protocols for a valid day of data will be used. Each parent with receive a logbook to complete each night to report non-wear time. Logs will be cross-referenced with the accelerometer data for quality assurance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Weaver RG, Armstrong B, Hunt E, Beets MW, Brazendale K, Dugger R, Turner-McGrievy G, Pate RR, Maydeu-Olivares A, Saelens B, Youngstedt SD. The impact of summer vacation on children's obesogenic behaviors and body mass index: a natural experiment. Int J Behav Nutr Phys Act. 2020 Nov 26;17(1):153. doi: 10.1186/s12966-020-01052-0. PMID 33243252